CLINICAL TRIAL: NCT06738810
Title: Identification of Non-alcoholic Steato-hepatitis Cases in a Sample of Type 2 Diabetes Patients, with a Disruption of the Liver Function Tests, At the Pointe-à-Pitre University Hospital
Brief Title: : Identification of Non-alcoholic Steato-hepatitis Cases in a Sample of Type 2 Diabetes Patients, with a Disruption of the Liver Function Tests, At the Pointe-à-Pitre University Hospital
Acronym: STEATOGWAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PAP_RI2_2017/06; 2017-A01101-52 (Other: ANSM)
Record Dates: First submitted 2022-07-01; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2022-07

CONDITIONS: Non-alcoholic Steato-hepatitis
Keywords: NASH,; type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: There will be a single group. Indeed, all type 2 diabetes with or without a hepatic check-up will be included in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- type 2 diabetes with a hepatic check-up patients (Other): For the study, a blood sample will be collected from the patient in order to do Fibrotest-actitest/NASHtest.
  Interventions: Diagnostic Test: Fibrotest-actitest/NASHtest

INTERVENTIONS:
Diagnostic Test: Fibrotest-actitest/NASHtest — A blood sample will be collected from the patient in order to do Fibrotest-actitest/NASHtest and to calculate the NAFLD fibrosis score
  Other Names: NAFLD fibrosis score

SUMMARY:
Non-alcoholic steatohepatitis (NASH) develops on insulin resistance, especially in patients with carbohydrate tolerance. NASH may progress to more extensive fibrosis, including cirrhosis, but also to HCC with or without cirrhosis in 10 to 20% of cases. The main objective of our research is to identify the prevalence of NASH in a sample of 100 patients with type 2 diabetes mellitus (T2DM), consulting in the PAP hospital and having a liver function disorder

DETAILED DESCRIPTION:
In Guadeloupe, the prevalence of T2DM is estimated to be 20%, among the highest in the French departements. NASH is probably present in our patients with T2DM but we do not know its prevalence. There is no data on the development of NASH in the Afro-Caribbean population, but in the United States, it has been observed that NASH was less prevalent among African-Americans compared to Caucasian and Hispanic Americans, and this could be explained by differences genetics in fat metabolism. In view of the emergence of NASH worldwide as a cause of chronic liver disease, it is necessary to carry out a pilot study to determine the presence or absence of NASH in T2DM patients in Guadeloupe. This will necessitate a systematic evaluation of liver function, usually performed during the T2DM assessment but not necessarily followed by specialized advice to confirm or invalidate the diagnosis of NASH. For each patient, an abnormality of liver function will be assessed by usual serum tests (transaminases, GGT, PAL). Prescription for a fibrotest / actitest + NASHtest and the NAFLD fibrosis score, will be perfomred as well as ultrasound and blood tests to eliminate other causes of liver disease (viral B or C, alcoholic, autoimmune, hemochromatosis) will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus patient with impaired hepatic function (transaminases and / or PAL and / or gamma-GT> Norm)
* Age ≥18 years
* Free, informed and written consent signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research).
* Affiliate or beneficiary of a social security scheme.

Exclusion Criteria:

* Pregnancy or breast-feeding
* No diabetes or type 1 diabetes
* Chronic hepatopathy of other origin: viral B, C, alcohol, hemochromatosis, α1-antitrypsin deficiency, Wilson's disease, autoimmune hepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
fibrotest-Actitest | 24 hours
  Fibrotest-actitest uses the biological analysis of alpha 2 macroglobulin, haptoglobin, apolipoprotein A1, total bilirubin, gGT, ALAT, ASAT, fasting blood glucose, cholesterol, triglycerides. A fibrotest score >0.48 is suggestive of advanced liver fibrosis.
NASH test | 24 hours
  NASHtest uses the biological analysis of alpha 2 macroglobulin, haptoglobin, apolipoprotein A1, total bilirubin, gGT, ALAT, ASAT, fasting blood glucose, cholesterol, triglycerides. NASHtest interpretation:
  NashTest 2 score Grade Interpretation
  0.00-0.25* N0 No NASH
  0.25-0.50* N1 Mild NASH
  0.50-0.75* N2 Moderate NASH
  0.75-1.00* N3 Severe NASH
NAFDL fibrosis score | 24 hours
  Non-Alcoholic Fatty Liver Disease (NAFLD) fibrosis score estimates amount of scarring in the liver based on age and body mass index of the patient, and several laboratory tests as ASAT, ALAT, platelet count and albumin. NAFLD fibrosis score can be interpretate as below:
  * less than -1.455: low probability of fibrosis
  * from -1.445 to 0.676 : intermediate score
  * more than 0.676: high probability of fibrosis

SECONDARY OUTCOMES:
: hepatic ultrasound, | 24 hours
  Patients will be assessed by liver ultrasound which is a non invasive test that produces images of liver and its blood vessels. It's a valuable diagnostic tool for assessing liver anatomy, size and pathology as cirrhosis or liver steatosis.
Standard liver test | 24 hours
  Blood analysis for liver function assessment (ASAT, ALAT, gGT, PAL)
Lipid balance | 24 hours
  Blood analysis for lipid metabolism assessment (total cholesterol, HDL cholesterol, triglycerides), which constitutes an important risk factor for cardiovascular disease
Lipid balance | 24 hours
  HDL
Lipid balance | 24 hours
  triglyceride
Assessment to eliminate other causes of chronic disease | 24 hours
  HBV and HCV serologies for viral hepatitis
Assessment to eliminate other causes of chronic disease | 24 hours
  auto-immune antibodies for auto-immune hepatitis
Assessment to eliminate other causes of chronic disease | 24 hours
  ferritinemia and saturation coefficient of transferin for hemochromatosis
Assessment to eliminate other causes of chronic disease | 24 hours
  carboxy deficient transferin for alcoholism
Platelets | 24 hours
  Platelet

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de la Guadeloupe, Pointe-à-Pitre, Pointe-à-Pitre, Guadeloupe

IPD SHARING:
Plan to Share IPD: No
Any plan has been do